CLINICAL TRIAL: NCT06524921
Title: Clinical and Radiographic Evaluation of Calcium Silicate Cement (Biodentine) Used As A Pulpotomy Agent In Primary Molars With Irreversible Pulpitis Versus Pulpectomy Using Calcium Hydroxide Iodoform Paste (Metapex)
Brief Title: Biodentine Pulpotomy vs Metapex Pulpectomy in Primary Molars: Clinical & Radiographic Comparison of Outcomes in Irreversible Pulpitis Cases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Ahmed Hamdi Abo El Yamin (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ahmed Hamdi Abo El Yamin, Dr., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-1
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: PICO:
  Population:
  Children with vital deeply carious primary molars with irreversible pulpitis
  Intervention:
  Pulpotomy using Biodentine in carious primary molars with irreversible pulpitis.
  Comparator/Control:
  Parial pulpectomy using Calcium Hydroxide with Iodoform ( Metapex ) in carious primary molars with irreversible pulpitis.
  Outcomes:
  Primary outcome, The presence of any adverse radiographic findings (Periodontal membrane space widening, periapical radiolucency, bone resorption, or other pathological changes)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metapex (Active Comparator): Partial pulpectomy using Calcium Hydroxide with Iodoform (Metapex ) in carious primary molars with irreversible pulpitis
  Interventions: Procedure: dental pulpectomy using metapex
- Biodentine (Experimental): Pulpotomy using Biodentine in carious primary molars with irreversible pulpitis
  Interventions: Procedure: dental pulpectomy using biodentine

INTERVENTIONS:
Procedure: dental pulpectomy using metapex — Metapex: A dental pulpectomy treats tooth with irreversible pulpitis in primary and teeth by removing infected pulp tissue using files and irrigation in the radicular part. The procedure involves anesthesia, decay removal, pulp chamber access, filing and irrigation till we reach cleaned dried canals and applying a medicament like Metapex . The tooth is then restored with a filling, often a stainless steel crown. The loss of pulp tissue weakens the tooth's structure and increases the risk of fracture and infection.
  Arms: Metapex
Procedure: dental pulpectomy using biodentine — Biodentine: A dental pulpotomy treats tooth decay or trauma in primary and young permanent teeth by removing infected pulp tissue in the crown while preserving healthy root pulp. The procedure involves anesthesia, decay removal, pulp chamber access, hemostasis, and applying a medicament like MTA or Biodentine. The tooth is then restored with a filling, often a stainless steel crown. Pulpotomies preserve tooth structure, relieve pain, and are less invasive than full root canals, but require regular follow-up.
  Arms: Biodentine

SUMMARY:
Irreversible pulpitis is defined as a clinical diagnostic based on subjective and objective findings suggesting that the vital inflamed pulp is incapable of healing in the American Association of Endodontists (AAE) Consensus Conference Recommended Diagnostic Terminology. Other characteristics include persistent heat discomfort, transferred pain, spontaneous pain, or no clinical symptoms but caries-induced inflammation, caries excavation, and trauma.".

Dental caries is one of the most frequently occurring diseases affecting human beings that becomes a challenge for dentists as the disease progresses. The ultimate goal of operative and endodontic treatment is to preserve and maintain the vitality of pulp to allow continued development of odontogenic apparatus.

DETAILED DESCRIPTION:
Pulp interventions combine a medication with a pulp treatment technique. Preserving the health of the tooth and its supporting tissues is the aim of these procedures. Three pulp therapy options are available, depending on the severity of the disease: pulpectomy, pulpotomy, and direct pulp capping. Direct pulp capping includes applying a medicinal material directly to the exposed pulp; pulpotomy and pulpectomy require removing parts of the pulp or the entire pulp in the pulp chamber and root canal of the tooth. In these procedures, the caries and part of pulp tissue are removed, and then medications are applied. This method aids in preserving the tooth's transient integrity.

When more advanced caries lesions approach the pulp-dentin complex and produce pulp necrosis, endodontic therapy is one way to save primary teeth until exfoliation. Maintaining the child's primary teeth in their oral cavity while getting rid of any symptoms or indicators is the ultimate goal of endodontic therapy in pediatric dentistry (Afroz et al., 2019).

zinc oxide eugenol (ZOE) was Introduced in 1930 and has been the conventional and widely approved root canal filling material for primary teeth. With over 90% of cases successfully reported, studies using ZOE paste have shown moderate to high success rates. But it has some drawbacks as well, such as the slower rate of resorption than the root, the possibility of the developing successor teeth becoming misaligned, particularly in overfilled cases, and worries about the material's potential for reduced antibacterial activity after the material is set in place.

Because zinc oxide eugenol has some disadvantages, biodentine-which may be utilized in direct contact with pulpal tissue-has strong mechanical properties, a good capacity to seal with dentine, and a biocompatibility that is comparable to that of MTA. It fulfilled every requirement of the perfect restorative material, including patient acceptance, good mechanical and physical properties, technical elements from the dentist's perspective, and other clinical characteristics that enhanced the material's efficacy. If only a portion of the odontoblastic layer is damaged, biodentine may accelerate pulp repair and regeneration.

For primary teeth pulpectomy, Metapex (Metapex, Meta Dental, New York, USA) is an easy-to-apply option that combines iodoform and calcium hydroxide. According to studies, this material has a good rate of resorption, less void formation, and excellent clinical and radiographic results.

ELIGIBILITY:
Inclusion Criteria:

* • Patient and parent showing cooperation and compliance.

  * Children 4-9 years old
  * Vital deeply carious primary(s) with complete root formation
  * Asymptomatic teeth or without clinical symptoms of spontaneous pain
  * No clinical evidence of pulp degeneration like the history of spontaneous or nocturnal pain, tenderness to percussion, pathologic tooth mobility, swelling, or fistulous tract.
  * Both genders will be included.
  * No radiographic evidence of pulp degeneration such as internal root resorption, external root resorption, or furcal radiolucency.
  * Presence of 2/3rd of root
  * Teeth that can be restored
  * Children with prior parental consent.

Exclusion Criteria:

* • soft tissue inflammation.

  * tooth mobility.
  * sinus tract.
  * Any radiographic sign of periapical pathologies or pulp necrosis (periapical radiolucency, internal or external root resorption)
  * History of any systemic disease
  * Teeth showing clinical or radiographic evidence of pulp degeneration
  * Hemostasis not achieved within 5 minutes of pulp amputation, by direct contact with a wet cotton pellet before the material placement
  * The remaining radicular tissue was non-vital (with suppuration or purulence necrosis)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic | Twelve Months
  Radiographic Furcation involvement: Furcation involvement will be assessed radiographically using DIGORA software, with visual interpretation assigning scores based on radiolucency levels: 0 for no radiolucency; 1 for radiolucency affecting up to ¼ of the furcation area extending towards the periapical region; 2 for radiolucency involving between ¼ and ½ of the furcation area extending towards the periapical region; and 3 for radiolucency affecting more than ½ of the furcation area extending towards the periapical region.

SECONDARY OUTCOMES:
Clinical | Twelve Months
  The presence of postoperative pain:The Wong-Baker FACES Pain Rating Scale, a self-report tool for acute pain, will be used to assess spontaneous pain and pain on biting. This scale ranges from 0 to 10, with six illustrated faces representing pain levels from "no hurt" to "hurts worst."

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salamoon, Ph.D, Study Chair — Lecturer of Pediatric Dentistry and Dental Public Health MSA University